CLINICAL TRIAL: NCT06149676
Title: A Novel Probiotic-antibiotic Combination to Prevent Recurrent Urinary Tract Infections
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Mehreen Arshad, Assistant Professor, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB 2022-4941
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Recurrent Uti
MeSH Terms: conditions — Urinary Tract Infections | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic with or without antibiotic (Experimental): All patients will receive probiotics for this, only those with a UTI will get ciprofloxacin.
  Interventions: Drug: Saccharomyces Boulardii 250 MG [Florastor]
- Control (No Intervention): Patients will get standard of care treatment.

INTERVENTIONS:
Drug: Saccharomyces Boulardii 250 MG [Florastor] — All patients will get the probiotic to be taken daily. If UTI occurs with a sensitive pathogen, we will treat with ciprofloxacin
  Other Names: ciprofloxacin
  Arms: Probiotic with or without antibiotic

SUMMARY:
Patients with recurrent UTI were randomized to receive either the probiotic Sacchromyces Boulardii at enrollment, and the intracellularly active Ciprofloxacin with their first UTI episode after enrollment, or they received standard of care treatment.

DETAILED DESCRIPTION:
* At the time of consent, participants will be given 20 mg/kg of the antibiotic, ciprofloxacin. If the participant has symptoms of a UTI or have a positive urine culture at enrollment, they will take the antibiotic every 12 hours for 14 days. If the participant does not have symptoms of a UTI at enrollment, the antibiotic will be taken only if needed at home upon the first occurrence of a UTI.
* At the time of consent, participants will also be given 250 mg of the probiotic, S.

boulardii, taken once daily for 6 months, irrespective of symptoms.

- Throughout the study, participants will receive their standard clinical care for recurrent UTI treatment, which includes bowel and bladder dysfunction management and other prescribed non-antibiotic interventions at the managing provider's clinical discretion.

ELIGIBILITY:
Inclusion Criteria:

* A history of 3 or more UTI episodes in the past 12 months, or 2 or more episodes in the past 6 months
* no evidence of vesicoureteral reflux or only low-grade (grade 1-2) vesicoureteral reflux
* no other genitourinary anatomical abnormality
* not receiving prophylactic antibiotics at the time of enrollment
* Ages 2-17 years.

Exclusion Criteria:

* high grade (grade 3-5) vesicoureteral reflux
* neurogenic bladder
* anatomical abnormalities of the gastrointestinal tract
* any history of urologic or gastrointestinal surgery
* on prophylactic antibiotics
* a urine culture positive for pathogens that are not susceptible to ciprofloxacin in the last 3 months
* history of an allergic reaction to ciprofloxacin or other quinolones, or a history of severe adverse reactions
* As stated on the package insert for Ciprofloxacin, individuals with a known history of myasthenia gravis should avoid taking Ciprofloxacin and therefore will be excluded from this study.
* Based on the black box warning for Ciprofloxacin, individuals taking tizanidine as concomitant administration, or those taking other drugs known to interact with ciprofloxacin will be excluded from the study.
* individuals with known QT prolongation, hypokalemia, or on other drugs that prolong the QT interval should also avoid taking Ciprofloxacin and will be excluded from this study.
* Individuals under 2 years old. In the BFIT clinic, because they do bladder, bowel movement, and constipation management, it is harder to manage if the patient is not potty trained. Therefore, we are excluding participants under 2 years of age.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in UTI episodes | 6 months
  We will look for a reduction the number of UTI episodes before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mehreen Arshad, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Lurie Children's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No